CLINICAL TRIAL: NCT06559475
Title: A Multicenter, Randomized Controlled Clinical Investigation to Evaluate the Safety and Effectiveness of the Super-Bore 8/7F Aspiration Catheters in the Treatment of Acute Intracranial Large Vessel Occlusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Super Aspiration
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke; Endovascular Thrombectomy
Keywords: Acute Ischemic Stroke; Super-Bore 8F Thrombosis Aspiration Catheter; Acute Intracranial Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super-Bore Thrombosis Aspiration Catheter treatment group (Experimental): For the subjects randomized to the Super-Bore Thrombosis Aspiration Catheter treatment group, mechanical thrombectomy will be performed using a Super-Bore 8/7F Thrombosis Aspiration Catheter.
  Interventions: Procedure: Super-Bore Thrombosis Aspiration Catheter treatment group
- Conventional thrombectomy device treatment group (Active Comparator): For the subjects randomized to the conventional thrombectomy device treatment group, mechanical thrombectomy will be performed using a commonly used thrombectomy devices in clinic, except for Super-Bore 8/7F Thrombosis Aspiration Catheter.
  Interventions: Procedure: Conventional thrombectomy device treatment group

INTERVENTIONS:
Procedure: Super-Bore Thrombosis Aspiration Catheter treatment group — For the subjects randomized to the Super-Bore Thrombosis Aspiration Catheter treatment group, Mechanical thrombectomy will be performed using a Super-Bore 8/7F Thrombosis Aspiration Catheter.
  Arms: Super-Bore Thrombosis Aspiration Catheter treatment group
Procedure: Conventional thrombectomy device treatment group — For the subjects randomized to the conventional thrombectomy device treatment group, mechanical thrombectomy will be performed using a commonly used thrombectomy devices in clinic, except for Super-Bore 8/7F Thrombosis Aspiration Catheter.
  Arms: Conventional thrombectomy device treatment group

SUMMARY:
To Evaluate the Safety and Efficacy of the Super-Bore 8/7F Thrombosis Aspiration Catheter in the Treatment of Acute Intracranial Large Vessel Occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Clinical presentation consistent with acute ischemic stroke (AIS);
3. Able to receive mechanical thrombectomy within 24 hours of onset;
4. Pre-morbid mRS score of 0 or 1;
5. Baseline NIHSS score of 6 or greater;
6. Complete or near-complete occlusion (eTICI 0-1) of the intracranial segment of the internal carotid artery (ICA), the M1 segment of the middle cerebral artery (MCA), or the basilar artery (with or without involvement of the intracranial vertebral artery) confirmed by angiography who can undergo intravascular thrombectomy;
7. Vessel diameter ≥2.2 mm at the occlusion site;
8. ASPECTS or PC-ASPECTS score of 6-10 on NCCT, CTA-source imaging, or DWI-MRI;
9. Written informed consent obtained from the patient or the patient's qualified representative.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Severe allergic reactions to contrast agents;
3. Current participation in other clinical studies;
4. Known hereditary or acquired bleeding disorders, platelet count <50,000/µL, or coagulation factor deficiencies;
5. Renal failure with serum creatinine ≥3 mg/dL or Glomerular Filtration Rate (GFR) <30 mL/min;
6. Expected survival < 6 months or known cancer with metastases;
7. Clinical manifestations suggesting subarachnoid hemorrhage, despite normal CT or MRI findings;
8. Suspected aortic dissection;
9. Known arterial condition in a proximal vessel that requires treatment or prevents access to the site of occlusion or safe recovery of the investigational device (for example, severe stenosis, complete occlusion in the cervical ICA, tandem occlusion);
10. High degree of suspicion of intracranial arterial disease (ICAD), such as evidence of multifocal ICAD on CTA, MRA, or DSA, or any other finding that is highly suggestive of ICAD as the underlying etiology of the occlusion;
11. Evidence of dissection in the extracranial or intracranial cerebral arteries;
12. Intracranial hemorrhage on CT or MRI;
13. Evidence of intracranial mass effect or tumor (except small meningiomas defined as ≤ 3cm and asymptomatic)) on CT or MRI;
14. Suspicious of cerebral vasculitis or infectious endocarditis;
15. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluation, e.g., dementia with prescribed anti-cholinesterase inhibitor;
16. Clinical history, past imaging or clinical judgement suggest that the intracranial occlusion is chronic;
17. Excessive vascular access tortuosity or target vessel size that will likely prevent endovascular access with the Super-Bore Aspiration Catheters;
18. Intracranial stent implanted in the same vascular territory that would preclude the safe deployment/removal of the thrombectomy devices;
19. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior circulation/vertebrobasilar system) as confirmed on CTA/MRA, or clinical evidence of bilateral strokes or strokes in multiple territories as determined by the treating physician;
20. Known aneurysm at or near the target treatment segment;
21. Known glucose level< 50 mg/dl (2.78 mmol/L) or > 400 mg/dl (22.20 mmol/L)；
22. Patients who, in the opinion of the investigator, are unsuitable for mechanical thrombectomy as evidenced by imaging findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The Rates of First Pass Effect (eTICI2c-3) | Within 5 minutes at final angiography of thrombectomy
  Evaluate effect of thrombectomy on reperfusion

SECONDARY OUTCOMES:
Proportion of mRS 0-2 at 90 days | 90 (± 14 days) after procedure
  Modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
90-day Global Disability Assessed Via the Blinded Evaluation of Modified Rankin Score (Ordinal Shift Analysis); | 90 (± 14 days) after procedure
  Modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

OTHER OUTCOMES:
Symptomatic intracerebral hemorrhage (sICH) | 24-48 hours after procedure
  sICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 24 hours , or any hemorrhage leading to death.
mortality | 90 (± 14 days) after procedure
  Number of subjects who died at 90-day follow-up/total number of subjects who participated in 90-day follow-up) x100%

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, MD, PhD, Study Chair — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No